CLINICAL TRIAL: NCT03030677
Title: Establishing Technique for PECS Type 2 (Serratus Block) Catheter Insertion With Ultrasound Guidence
Brief Title: Establishing Technique for PECS2 Catheter Insertion
Acronym: ETCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mansour, assistant professor, anesthesia department, kasr al aini faculty of medicine, cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MMSTD1Pecs2
Record Dates: First submitted 2017-01-05; First posted 2017-01-25 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Breastcancer; Phyllodes Breast Tumor
Keywords: pecs block; breast surgery; ultrasound guidence
MeSH Terms: conditions — Phyllodes Tumor | interventions — Catheters; Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Without Dissectioin (Other): confirming insertion of B Braun Catheter Kit Contiplex with 18 Gauge needle using ultrasound without injecting 10 ml of lidocaine 1% as a dissecting solution
  Interventions: Procedure: Pectoralis II block & catheter without Lidocaine dissection; Other: catheter insertion
- Interventional With Dissectioin (Other): confirming insertion of B Braun Catheter Kit Contiplex with 18 Gauge needle using ultrasound after injecting 10 ml of lidocaine 1% as a dissecting solution
  Interventions: Procedure: Pectoralis II block & catheter with Lidocaine dissection; Other: catheter insertion

INTERVENTIONS:
Procedure: Pectoralis II block & catheter without Lidocaine dissection — B Braun Catheter Kit Contiplex with a 18 gauge needle will be used. After topicalization of the skin and sterilization using ultrasound guidance to facilitate performing insertion of the canula. Confirming the tip position will be done by ultrasonography while performing pectoralis type 2 block for cases undergoing simple mastectomy procedures
  Arms: Interventional Without Dissectioin
Procedure: Pectoralis II block & catheter with Lidocaine dissection — B Braun Catheter Kit Contiplex with a 18 gauge needle will be used. After topicalization of the skin and sterilization using ultrasound guidance to facilitate performing insertion of the canula. 10 ml of lidocaine 1% will be injected for plan dissection to facilitate the procedure. Confirming the tip position will be done by ultrasonography while performing pectoralis type 2 block for cases undergoing simple mastectomy procedures
  Arms: Interventional With Dissectioin
Other: catheter insertion — catheter insertion after Lidocaine dissection

SUMMARY:
The investigators are trying to establish an easy technique for insertion of a catheter for continuous infusion while performing pectoral type 2 (serratus) block, as a post operative pain controlling measure for cases undergoing simple mastectomy, using ultrasound guidence

DETAILED DESCRIPTION:
As the space between the pectoralis minor and the serratus anterior is a fashial plane with a connective tissue occupying. we are trying to demonstrate a simple technique for inserting a catheter within that fashial plane and making sure of the catheter position, to ensure post operative analgesia for cases performing simple mastectomy.

Now the Pectoralis type 2 block (PECS type 2) is an established technique as regional block technique for chest wall procedures.

We are trying to maximizing the benefit of the block with a catheter insertion to use it for continuous infusion of bupivacaine for controlling post operative pain in cases performing simple mastectomy procedure

ELIGIBILITY:
Inclusion Criteria:

* Female patient scheduled for simple mastectomy
* Accepted performing the block

Exclusion Criteria:

* Patients on anticogulants
* Chest wall infection
* Patient refusal

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
successful catheter insertion | during time of performing the block
  confirming catheter insertion 5 cm beyond the tip of needle in the proper plan using ultrasound

SECONDARY OUTCOMES:
Number of attempts | during time of performing the block
  Number of attempts needed for successful insertion
Duration needed for insertion | during time of performing the block
  Duration needed for successful insertion

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ah Mansour, ass.prof, Principal Investigator — Kasr Al Aini Faculty of Medicine
Locations (1):
- Kasr Alaini Hospitals, Cairo, Egypt

REFERENCES:
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/27871558